CLINICAL TRIAL: NCT06300437
Title: The Effects of Jaw Thrust on the Time to Successful Fiberoptic Pediatric Orotracheal Intubation During Residents Training Program, a Randomized Controlled Trial
Brief Title: The Effects of Jaw Thrust on the Time to Successful Fiberoptic Pediatric Orotracheal Intubation During Residents Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-372-2023
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Intubation
Keywords: fiberoptic; intubation; children; training

STUDY DESIGN:
Intervention Model Description: In this study, children undergoing elective surgery under general anesthesia will be randomized into 2 groups.
  * Group (J): will include the children who will receive jaw thrusting during fiberoptic intubation.
  * Group (C): will include the children who will not receive jaw thrusting (just sub laxed open mouth)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group jaw thrust (Experimental): will include the children who will receive jaw thrusting during fiberoptic intubation.
  Interventions: Procedure: jaw thrust
- Group control (Active Comparator): will include the children who will not receive jaw thrusting (just sub laxed open mouth)
  Interventions: Procedure: control (sub laxed jaw)

INTERVENTIONS:
Procedure: jaw thrust — children who will receive jaw thrusting during fiberoptic intubation
  Arms: Group jaw thrust
Procedure: control (sub laxed jaw) — children who will not receive jaw thrusting (just sub laxed open mouth)
  Arms: Group control

SUMMARY:
In this study, the authors aim to investigate the effect of adding jaw thrust maneuver on time to successful orotracheal fiberoptic intubation of pediatrics during resident training program.

DETAILED DESCRIPTION:
In this study, children undergoing elective surgery under general anesthesia will be randomized into 2 groups.

* Group (J): will include the children who will receive jaw thrusting during fiberoptic intubation.
* Group (C): will include the children who will not receive jaw thrusting (just sub laxed open mouth) Following approval from the Research and Ethics Committee of the anesthesia department, Faculty of Medicine, Cairo University, and obtaining written informed consent from all participating children parents' meeting the inclusion criteria; children will be randomly assigned into two groups using a computer-generated random number list with a closed-sealed envelope.
* Group (J): will include the children who will receive jaw thrusting during fiberoptic intubation.
* Group (C): will include the children who will not receive jaw thrusting (just sub laxed open mouth) The day before the operation, all children guardians' will be instructed to follow institutional fasting guidelines (a minimum of 2 h for clear fluids, 4 h for breast milk, and 6 h for formula feeding or light meals).

All children will receive an inhalation induction with sevoflurane in oxygen 100% and will be monitored with pulse oximetry, noninvasive blood pressure monitoring, electrocardiography, and end-tidal carbon dioxide monitoring. An intravenous line will be inserted, Atropine 0.01mg/kg with a minimum of 0.1mg will be given and anesthesia will be completed with 1µ/kg fentanyl and 0.5 mg/kg Atracurium. Children will then be preoxygenated using appropriate mask and volume-controlled ventilation (VCV) using (G.E-Datex-Ohmeda, Avance CS2, USA). Ventilation will be set at 6 ml/kg, respiratory rate of 20 and PEEP 3 cmH2O with 100% O2, and 2% sevoflurane for at least 3 min before intubation attempts. Adequate ventilation will be ensured using end-tidal carbon dioxide monitoring. At least 4 randomly selected residents will participate in the study. The residents performing the fiberoptic intubations will not be involved in induction of anesthesia for the children. Each resident had completed at least 2 years of anesthesia residency training program and had at least 5 fiberoptic intubation on mannequin under supervision of the airway management committee members in Kasr Alainy, Cairo University. All residents will receive the same orientation to using fiberscopes in children before their first intubation attempt. Each resident will attempt fiberoptic intubation in at least 10 patients in each group randomly under direct guidance of the same attending senior anesthesiologist. The fiberoptic (Storz ®Flexible intubation video endoscope (FIVE) 4.0 mmx65cm attached to the multifunctional C-MAC® monitor) will be prepared by an anesthesia nurse using an antifogging solution and a suction catheter will be applied to the suction channel and connected to the wall vacuum. All endotracheal tubes will be loaded onto the fiberscope with the Murphy eye up (bevel facing down) which will be kept in position using adhesive tape throughout the whole procedure to facilitate successful placement of endotracheal tube into the trachea. The supervising anesthesiologist (not blinded to the assigned group) will secure the child's head in a neutral position and held the mouth open and the jaw sub laxed while providing verbal instruction to the assigned resident in the controlled group while in the jaw thrust group the supervising anesthesiologist will maintain the jaw thrusted while giving instruction to the training resident by placing the index and middle fingers to push the posterior aspects of the lower jaw upwards while his thumbs push down on the chin to open the mouth. Instruction for the residents will be based on the shared view of the airway on the fiberoptic screen during the course of intubation. During intubation, the anesthesia nurse will use a stopwatch to measure the duration of each intubation attempt and the time from mask removal to confirmation of endotracheal tube placement by direct visualization of the ETT in the trachea. An intubation attempt will be aborted if there is a decrease in oxygen saturation to 93% before completion of intubation or if the attempt takes longer than 3 min. The patients will be ventilated with 100% O2 and 3% sevoflurane for 3 min between attempts. Three attempts will be permitted for fiberoptic intubation. If 3 attempts for fiberoptic intubation failed, the child will be intubated using direct laryngoscope and the child will be excluded from the study. The number of attempts required for successful completion of intubation will be recorded, the failure rate and the cause of failure (failure to correctly place the fiberscope or failure to thread the endotracheal tube into the trachea) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children more than 1-year of age
* American Society of Anesthesiologists physical status I-II
* scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* Patients known or suspected difficult intubation.
* Patients with syndrome known to be associated with difficult intubation.
* Patients with severe pulmonary or cardiac diseases.
* Patients at risk of aspiration (patients with lower esophageal disease such as Hiatus hernia, or GERD and DM).
* Body mass index (BMI) greater than 35 kg/m2.
* Refusal of the patient guardians.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
time to successful endotracheal tube insertion | 3 minutes
  time to successful endotracheal tube insertion (defined as time from face mask removal until direct visualization of the ETT in the trachea by the fiberscope after sliding of the ETT over the fiberscope).

SECONDARY OUTCOMES:
Number of attempts to successful intubation | 3 minutes
  Number of attempts to successful intubation
Complication | 3 minutes
  example: airway trauma, severe desaturation SPO2 below 90%

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No